CLINICAL TRIAL: NCT04505163
Title: Left Atrial Posterior Wall Isolation in Conjunction With Pulmonary Vein Isolation Using the Cryoballoon for Treatment of Persistent Atrial Fibrillation (PIVoTAL) - IDE Trial
Brief Title: Left Atrial Posterior Wall and PV Isolation Using Cryoballoon for Treatment of Persistent AF
Acronym: PIVoTAL-IDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dignity Health Medical Foundation (Other)
Collaborators: Mercy General Hospital and Dignity Health Medical Foundation (Unknown); Beth Israel Deaconess Medical Center (Other); UC Health Medical Center (Unknown); MedStar Georgetown University Hospital and Medical Center (Unknown); Tampa Cardiac Specialists (Unknown); Bethesda North Hospital (Unknown); Brigham and Women's Hospital (Other); Texas Cardiac Arrhythmia Institute At St. Davids Medical Center (Unknown); St. Luke's Hospital and Health Network, Pennsylvania (Other); Sarasota Memorial Health Care System (Other); Nebraska Methodist Hospital-Methodist Physicians Clinic (Unknown)
Responsible Party: Principal Investigator, Arash Aryana, MD, Principal Investigator, Dignity Health Medical Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIVoTAL-IDE
Record Dates: First submitted 2020-07-10; First posted 2020-08-10 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Catheter ablation; Cryoablation; Cryoballoon; Posterior left atrial wall ablation; Pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Cryoballoon Pulmonary Vein Isolation (PVI) (Active Comparator): Standard cryoballoon pulmonary vein isolation alone using the Arctic Front Advance Cryoablation System family of cardiac ablation catheters
  Interventions: Procedure: Standard Cryoballoon Pulmonary Vein Isolation (PVI)
- Cryoballoon PVI + Posterior Wall Isolation (Experimental): Cryoballoon pulmonary vein isolation in conjunction with posterior wall isolation using the Arctic Front Advance Cryoablation System family of cardiac ablation catheters
  Interventions: Device: Cryoballoon PVI + Posterior Wall Isolation

INTERVENTIONS:
Procedure: Standard Cryoballoon Pulmonary Vein Isolation (PVI) — Arctic Front Advance cryoballoon ablation system to ablate the pulmonary veins to achieve PVI alone
  Other Names: Arctic Front Advance Cardiac Cryoablation System
  Arms: Standard Cryoballoon Pulmonary Vein Isolation (PVI)
Device: Cryoballoon PVI + Posterior Wall Isolation — Arctic Front Advance Cardiac Cryoballoon Ablation System to ablate the pulmonary veins and the left atrial posterior wall to achieve PVI + posterior wall isolation within the region of the pulmonary venous component
  Other Names: Arctic Front Advance Cardiac Cryoablation System
  Arms: Cryoballoon PVI + Posterior Wall Isolation

SUMMARY:
The purpose of this study it to learn whether pulmonary vein isolation (PVI) along with isolation of the posterior left atrial wall (PWI) in the region of the pulmonary venous component will reduce the likelihood of atrial fibrillation (AF) recurrence in patients with persistent atrial fibrillation at 12 months, after a single ablation procedure, in comparison to PVI alone.

The investigator hypothesizes that the combination of PVI + PWI will result in a significant reduction in recurrence of atrial fibrillation at 12 months after ablation.

DETAILED DESCRIPTION:
Patients with persistent atrial fibrillation will be enrolled in this multi-center, randomized, prospective, single-blinded study. After catheter ablation (isolation) of the pulmonary veins (PVI) and while still in the cardiac electrophysiology laboratory, all patients will be randomized to either PVI alone or the combination of PVI + posterior left atrial wall isolation (PWI). For patients randomized to PVI, their ablation procedure will be completed at that time. For those patients randomized to PVI + PWI, they will have additional ablation to achieve PWI.

All study patients will have the same follow-up after their ablation procedure, including clinic visits at 3, 6, and 12 months and a heart event monitor for 7-14 days before these visits. An echocardiogram (heart ultrasound) is performed at 6 to 12 months after the ablation. Blood thinners are recommended for two months after ablation and then the need for continued use of blood thinners will be based on individual patient's medical history, stroke risk and the decision of the study doctor. Information about the patients' medical history, heart arrhythmias and atrial fibrillation will be collected during the study which will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Consistent with the current definitions, all patients with Persistent AF must exhibit an episode of continuous AF that is sustained >7 days.
* Patients must have symptomatic Persistent AF refractory or intolerant to at least one class I or class III antiarrhythmic drug
* Males and females with an age >18 years undergoing a first-time catheter ablation of AF; prior ablation of a right atrial cardiac arrhythmia (i.e., typical right atrial flutter) is permitted
* All patients must understand the requirements of the study and be willing to comply with the post-study follow-up requirements
* Patients must have documented episode of AF greater than 7 days in the year prior to the procedure

Exclusion Criteria:

* History of long-standing persistent AF
* Any reversible cause of AF (post-operative, thyroid disorder, etc.)
* Patients with cerebral ischemic events (stroke or transient ischemic attack), myocardial infarction or unstable angina in the previous 2 months
* Patients with any corrected or uncorrected congenital heart disease
* Patients with a history of hypertrophic cardiomyopathy
* Patients with cardiomyopathy and a left ventricular ejection fraction <40%
* Congestive heart failure, class IV
* Left atrial (LA) diameter >55 mm (parasternal long axis view)
* Patients with left atrial thrombus
* Women who are known to be pregnant or have had a positive β-HCG (human chorionic gonadotropin) test 7 days prior to procedure
* Patients whose life expectancy is <1 year
* History of left-sided left atrial ablation (catheter or surgically-based)
* Mental impairment precluding the patient from providing informed consent or completing appropriate follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
12-month freedom from recurrent atrial fibrillation | 12 months
  Number of participants with recurrent atrial fibrillation following catheter ablation

SECONDARY OUTCOMES:
All atrial arrhythmia recurrences | During a follow-up period of 12 months
  Number of atrial arrhythmia recurrences after the 90-day blanking period
Change in Canadian Cardiovascular Society Severity of Atrial Fibrillation Scale (CCS-SAF) | During a follow-up period of 12 months
  Change in CCS-SAF from baseline to 12 months
Change in Atrial Fibrillation Effect on Quality of Life Questionnaire (AFEQT) | During a follow-up period of 12 months
  Change in AFEQT from baseline to 12 months
Multiple procedure success | During a follow-up period of 12 months
  Absence of recurrent atrial arrhythmias after one or more ablation procedure(s)
Relative reduction in atrial fibrillation burden | During a follow-up period of 12 months
  Reduction in the burden of atrial fibrillation (in percentage) following catheter ablation
Freedom from cardioversion for recurrent atrial arrhythmias | During a follow-up period of 12 months
  Electrical or pharmacological cardioversion for treatment of recurrent atrial arrhythmias not required
Freedom from repeat atrial fibrillation ablation | During a follow-up period of 12 months
  Repeat ablation for atrial fibrillation
Left Atrial Diameter (Size) as predictor of atrial fibrillation recurrence | During a follow-up period of 12 months
  Change in left atrial diameter (in millimeters) following ablation
Left Ventricular Ejection Fraction as predictor of atrial fibrillation recurrence | During a follow-up period of 12 months
  Change in left atrial ejection fraction (in percentage) following ablation
New York Heart Association Functional Class as predictor of atrial fibrillation recurrence | During a follow-up period of 12 months
  Change in New York Heart Association Functional Class following ablation

CONTACTS AND LOCATIONS:
Overall Officials: Arash Aryana, MD, Principal Investigator — Mercy General Hospital and Dignity Health Medical Foundation
Locations (11):
- United States (11):
  - Mercy General Hospital and Dignity Health Medical Foundation, Sacramento, California
  - UCHealth Medical Center, Fort Collins, Colorado
  - MedStar Georgetown University Hospital and Medical Center, Washington D.C., District of Columbia
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Tampa Cardiac Specialists, Tampa, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Nebraska Methodist Hospital-Methodist Physicians Clinic, Omaha, Nebraska
  - Bethesda North Hospital, Cincinnati, Ohio
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Texas Cardiac Arrhythmia Institute & St. David's Medical Center, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aryana A, Pujara DK, Allen SL, Baker JH, Espinosa MA, Buch EF, Srivatsa U, Ellis E, Makati K, Kowalski M, Lee S, Tadros T, Baykaner T, Al-Ahmad A, d'Avila A, Di Biase L, Okishige K, Natale A. Left atrial posterior wall isolation in conjunction with pulmonary vein isolation using cryoballoon for treatment of persistent atrial fibrillation (PIVoTAL): study rationale and design. J Interv Card Electrophysiol. 2021 Oct;62(1):187-198. doi: 10.1007/s10840-020-00885-w. Epub 2020 Oct 3. PMID 33009645